CLINICAL TRIAL: NCT04663061
Title: Data-Assisted Approach for High Intensity Medical Weight Loss for Diabetes Remission
Brief Title: Diabetes Data-Assisted Remission Trial (DDART)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: UnitedHealth Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00067950
Record Dates: First submitted 2020-12-09; First posted 2020-12-10 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes; Obesity
Keywords: Diabetes; Obesity; Weight management; Diabetes education; Diabetes remission
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High intensity medical weight loss (HIWL) (Experimental): Participants randomized to the HIWL treatment group will be placed on a meal replacement-based weight loss protocol. Participants will consume a minimum of 80 grams of protein daily in 4-5 servings of meal replacement. Participants will begin to incorporate food into their routine beginning at week 13 with guidance from a dietitian. From weeks 13-24, caloric prescriptions will be between 1100 to 1600 calories a day, using a combination of meal replacements and food, for continued weight loss. Beyond week 25, caloric intake will be individually tailored to achieve continued gradual weight loss or maintenance of body weight based on individual weight loss goals. We will recommend continued use of at least 1 serving of meal replacement per day for maintenance of weight loss.
  Interventions: Behavioral: Medical weight loss
- Diabetes self-management education (DSME) (Active Comparator): The DSME intervention will be administered and delivered at the Wake Forest Baptist Health Diabetes Center, located next to the Weight Management Center, by a team of certified diabetes educators, nurses, and nutritionists in group and individual settings.
  The diabetes education program is accredited by the American Diabetes Association in recognition of meeting national standards for diabetes self-management education. The goal of the program is to provide participants with information to make informed decisions about how to best integrate diabetes management strategies into their daily lives. Assessment, planning, implementation, and evaluation are the basic components of the diabetes education process.
  Interventions: Behavioral: Diabetes education
- High intensity medical weight loss (HIWL) plus continuous glucose monitoring (CGM) (Experimental): Participants randomized to the HIWL + CGM treatment group will be placed on a meal replacement-based weight loss protocol as described in the HIWL arm. In addition, the participants in this arm will receive a supply of continuous glucose monitors to use throughout the trial. The CGM we provide will give the patient instant feedback on blood glucose levels and be readable using a mobile phone device or an associated CGM reader. The data from the CGM will be integrated into the Carium app and used to help guide the patient's actions based on defined care pathways.
  Interventions: Behavioral: Medical weight loss; Behavioral: Continuous glucose monitoring

INTERVENTIONS:
Behavioral: Medical weight loss — Participants will be prescribed intensive medical weight loss with the goal of achieving 15% weight loss from initial weight
  Arms: High intensity medical weight loss (HIWL); High intensity medical weight loss (HIWL) plus continuous glucose monitoring (CGM)
Behavioral: Diabetes education — Participants will receive standard of care diabetes education
  Arms: Diabetes self-management education (DSME)
Behavioral: Continuous glucose monitoring — Participants will use CGM devices to track blood glucose levels in near real time
  Arms: High intensity medical weight loss (HIWL) plus continuous glucose monitoring (CGM)

SUMMARY:
The study team will study the efficacy of a high intensity medical weight loss intervention paired with a digital platform to create weight loss and induce remission of type 2 diabetes mellitus (T2DM) compared to a diabetes self-management education intervention. The digital platform provides the capability to tailor the treatment plan, provide automated support, and alert providers when a participant may need more support from the clinical team. If shown to be efficacious, this research could be highly impactful, causing us to rethink our approach to care for those with T2DM and shift the paradigm for millions of individuals in the United States. Furthermore, this approach will demonstrate the feasibility of helping people engage in metabolic treatment strategies in a way that is scalable leveraging digital and mobile solutions that extend the patient-provider relationship, shift care from episodic approaches to more of an on-going model that extends into the life of the patient, while also integrated within the healthcare system workflows.

DETAILED DESCRIPTION:
This project will determine if a data-assisted, high intensity medical weight loss intervention (HIWL) will lead to significant weight loss and diabetes remission in individuals with a Body Mass Index (BMI) 30-39.9 kg/m2 with T2DM of less than 6 years as compared to a diabetes self-management education intervention (DSME). Complete diabetes remission is considered to be achieved when the patient is not taking any anti-diabetes medication for at least 12 months, and the Glycated Hemoglobin (HbA1c) is < 5.7%. Partial remission is achieved when the patient is not taking any anti-diabetes medication and has an HbA1c of 5.7-6.4% for at least 12 months.Using a randomized controlled study design, we will randomly assign 90 participants to HIWL, HIWL + continuous glucose monitoring (CGM), or DSME. Participants assigned to HIWL will receive a high intensity behavioral weight loss intervention delivered using a digital patient engagement platform. Participants will be prescribed a low calorie dietary plan and a recommended physical activity program designed to produce 15-20% weight loss over 12 months. Those assigned to HIWL + CGM will receive the same intervention as HIWL; in addition we will provide them with CGM to use as part of their remote monitoring on a daily basis. Those assigned to DSME will participate in a comprehensive diabetes education program designed to provide education and skills for optimal diabetes management plus lifestyle modification counseling to produce 5% weight loss over the same timeframe. The primary outcome of weight loss will be assessed at 12 months.

ELIGIBILITY:
Inclusion:

* Individuals with T2DM diagnosed within the past 6 years
* Body Mass Index (BMI) of 30-39.9 kg/m2.
* Participants must have an HbA1c between 6.5-11.9%.
* Participants should be able to participate in all aspects of the recommended interventions, including being able to participate in exercise, make recommended dietary changes, and engage in individual and group counseling.

Exclusion criteria:

* Poorly controlled depression
* Recent hospitalization for psychosis or bipolar disorder
* Poorly controlled blood pressure (>159/99)
* Prior surgical procedure for weight control or liposuction
* Unable to make changes to their diet
* Unable to exercise (walk for at least 6 minutes and perform simple strength and stretch exercise tests)
* Use of weight loss medications in previous 3 months
* Recent self-reported weight change (+/- 15lbs)
* Current use of oral corticosteroids more than 5days/month
* Cardiovascular disease event within the past 6 months
* Severe pulmonary disease requiring supplemental oxygen
* Renal failure (end stage renal disease)
* History of non-skin cancer in the past 5 years
* Major liver dysfunction within the last 2 years
* Recently quit smoking less than 6 months prior
* Inability to attend visits and adhere to study protocols
* Pregnancy or currently lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2024-11-14 (Actual); Study Completion 2024-11-14 (Actual)

PRIMARY OUTCOMES:
Change in Body Weight | baseline through 12 months
  Change in weight from baseline

SECONDARY OUTCOMES:
Change in Hemoglobin A1c | baseline through 12 months
  Change in hemoglobin A1c
Number of Subjects in Diabetes Remission | 12 months
  Achieving A1c <6.5% and no anti-diabetes medications
Continuous Glucose Monitoring (CGM) Time in Range | baseline through 12 months
  Collected by FreeStyle Libre. Average time spent at an average glucose of 100 mg/dL or lower.
CGM Time in Range--Post-meal Glucose | baseline through 12 months
  Collected by FreeStyle Libre. Average time spent at a post-meal glucose level of 110 mg/dL or lower.
CGM Time in Range--Fasting Glucose | baseline through 12 months
  Collected by FreeStyle Libre. Average time spent in normal fasting glucose between 72-85 mg/dL.
CGM Episodes of Hypoglycemia | baseline through 12 months
  Collected by FreeStyle Libre. Number of episodes.
CGM Glucose Variability | baseline through 12 months
  Collected by FreeStyle Libre. Coefficient of variance
CGM Average Glucose | baseline through 12 months
  Collected by FreeStyle Libre.
Automated Self-Administered 24-hour (ASA24) Total Daily Energy Intake | baseline, 3 months, 6 months, and 12 months
  kilocalories averaged across 3 days
ASA24 Macronutrient Composition of Diet | baseline, 3 months, 6 months, and 12 months
  %Carbohydrate/Fat/Protein; averaged across 3 days
ASA24 Number of Eating Episodes Per Day | baseline, 3 months, 6 months, and 12 months
  averaged across 3 days
ASA24 Healthy Eating Index (HEI)-2015 score | baseline, 3 months, 6 months, and 12 months
  A validated summary measure of dietary quality, rated on a 100-point scale with a higher score denoting better diet quality
Daily Step Counts | baseline, 3 months, 6 months, and 12 months
  Collected by pedometer over 7 days during each period. At the end of the 7th day, participants will record the final step count, and return the pedometer to the study team via a pre-stamped mail envelope.
International Physical Activity Questionnaire (IPAC) short form: moderate-vigorous physical activity minutes | baseline, 3 months, 6 months, and 12 months
  A validated self-report measure of daily physical activity levels. Responses are given as minutes per day over the last week of moderate and vigorous physical activity. Outcome is average total minutes/week.
International Physical Activity Questionnaire (IPAC) short form: walking minutes | baseline, 3 months, 6 months, and 12 months
  A validated self-report measure of daily physical activity levels. Responses are given as minutes per day over the last week of walking for exercise. Outcome is average total minutes/week.
International Physical Activity Questionnaire (IPAC) short form: sitting time | baseline, 3 months, 6 months, and 12 months
  A validated self-report measure of daily physical activity levels. Responses are given as minutes per day over the last week of sitting time. Outcome is average total minutes/week.

CONTACTS AND LOCATIONS:
Overall Officials: Jamy Ard, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Univesity Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results of any reported manuscripts after deidentification will be made available for the specified timeframes. Researchers who provide a methodologically sound proposal for analysis will be granted access.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following any publication.
Access Criteria: Proposals will need to be sent to jard@wakehealth.edu for review and approval. To gain access, data requestors will need to sign a data access agreement.

DOCUMENTS (1):
  • Informed Consent Form (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT04663061/ICF_000.pdf